CLINICAL TRIAL: NCT06826196
Title: A Phase 1B/2A, Randomized, Double-blind, Placebo-controlled, Intraindividual Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of ALD-102 Solution in Subjects With Alopecia Areata
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of ALD-102 Solution in Subjects With Alopecia Areata
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aldena Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ALD-102Sol-001
Record Dates: First submitted 2025-01-22; First posted 2025-02-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Alopecia Areata (AA)
MeSH Terms: conditions — Alopecia Areata | interventions — reproxalap

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- ALD-102 (Experimental)
  Interventions: Drug: ALD-102

INTERVENTIONS:
Drug: ALD-102 — Treatment every 4 weeks for total of 8-week treatment period.
  Arms: ALD-102
Drug: Placebo — Treatment every 4 weeks for 8-week treatment period
  Arms: Placebo

SUMMARY:
The goal of this first-in-human clinical trial is to learn if ALD-102 Solution is safe and well tolerated following injections in the scalp in subjects with alopecia areata. The study will also learn about the effect of ALD-102 on hair regrowth in treatment areas. The researchers will compare the effects of ALD-102 Solution (drug) to placebo (saline solution that contains no drug). Study participants will have two treatment areas selected on the scalp and will receive randomly ALD-102 Solution (drug) at one area and or placebo (saline solution) at the other area once every 4 weeks for a treatment period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged 18 to 55 years, inclusive, at the time of informed consent.
2. Subject has a body mass index (BMI) between 18.0-35.0 kg/m2, inclusive, at screening.
3. Subject has a body weight ≥ 50 kg, inclusive, at screening.
4. Subject has a clinically confirmed diagnosis of AA at screening visit, based on investigator's judgement.
5. Subjects with AA lesion(s) that can accommodate for 2 separate treatment areas large enough to receive 20 injections each (Cohort 1) or to receive 40 injections each (Cohorts 2-4). The 2 treatment areas must be clinically similar as per investigator's judgment, ≥ 6 cm apart, and can be located on the same AA lesion or on 2 different AA lesions.
6. Duration of current episode of hair loss at the treatment areas > 6 months but < 5 years at screening and Day 1, along with investigators' assessment that hair regrowth is possible. Total duration of current episode of hair loss outside of treatment areas and total duration since diagnosis of AA could be > 5 years.
7. No evidence of active regrowth or hair loss present at baseline and no known history of significant regrowth or hair loss, as per investigator's judgement, over the last 6 months.
8. Subject is willing to keep the same hairstyle and color (eg, hair products, process, and timing for hair appointments) for the duration of the trial.

   Note: Hair dying and shaving of scalp is allowed during the trial but not within 2 weeks prior to a study visit.
9. For female subject of childbearing potential involved in any sexual intercourse that could lead to pregnancy: the subject must agree to use a highly effective contraceptive method in addition to use of condom for their non-vasectomized male partner(s) from ≥ 4 weeks prior to Day 1 until ≥ 16 weeks after the last injection, and refrain from egg retrieval/egg donation during this period. Highly effective contraceptive methods include hormonal contraceptives (eg, combined oral contraceptive, patch, vaginal ring, injectable, or implant), intrauterine devices or intrauterine systems, vasectomized partner(s) (provided his vasectomy was performed ≥ 4 months prior to Screening), tubal ligation or double barrier methods of contraception (eg, male condom with cervical cap, male condom with diaphragm, and male condom with contraceptive sponge) in conjunction with spermicide.

   Note: Subjects must have been on a stable dose of hormonal contraceptives for ≥ 4 weeks before Day 1.

   Note: The above list of contraceptive methods does not apply to subjects who are abstinent for ≥ 4 weeks before Day 1 and will continue to be abstinent from penile-vaginal intercourse throughout the trial or for ≥ 16 weeks after the last injection. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not acceptable.

   Note: A female subject of nonchildbearing potential is defined as follows:
   * Female subject who has had surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy)
   * Female subject who has had a cessation of menses for ≥ 12 months prior to the screening visit without an alternative medical cause, and a follicle-stimulating hormone (FSH) test confirming nonchildbearing potential (refer to laboratory reference ranges for confirmatory levels).
10. For male subject involved in any sexual intercourse that could lead to pregnancy, subject must agree to use a condom and their female partner must use one of the highly effective contraceptive methods listed in Inclusion Criterion #9, from Day 1 until ≥ 16 weeks after the last injection and refrain from donating sperm during this period. If the female partner of a male subject uses any of the hormonal contraceptive methods listed above, this contraceptive method should be used by the female partner from ≥ 4 weeks before Day 1 until ≥ 16 weeks after the last injection.
11. Female subject of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test at Day 1.
12. Subject is willing to participate and is capable of giving a signed and dated informed consent.

    Note: Consent must be obtained prior to any study-related procedures.
13. Subjects must be willing to comply with all study procedures and must be available for the duration of the study.
14. Subjects must be willing to receive between approximately 40 to 80 intradermal injections every 4 weeks (number of injections will vary for each cohort).

Exclusion Criteria:

1. Very severe AA, defined by SALT score ≥ 95 at screening and/or Day 1, including alopecia universalis and alopecia totalis.
2. Presence of another form of alopecia (eg, androgenetic alopecia, traction and scarring alopecia, telogen effluvium).
3. Presence of diffuse type of AA, or presence of ophiasis or sisapho patterns of AA.
4. History or presence of hair transplants.
5. History or presence of micropigmentation of the scalp. Note: microblading of the eyebrows is permitted.
6. Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
7. Subject is known to have immune deficiency or is immunocompromised.
8. Subject has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1. Subjects with successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded.
9. Subject had a major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
10. Subject has any clinically significant medical condition or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with the interpretation of trial results.
11. Subject has a positive result for hepatitis B virus (HBV; positive for hepatitis B surface antigens [HBsAg] or positive for hepatitis B antibodies to core antigens [anti-HBc]; subjects having a negative HBsAg and a positive anti-HBc may enroll if they have a positive hepatitis B surface antibody [anti-HBs] demonstrating natural immunity), hepatitis C virus (HCV; positive for HCV antibodies; however, a subject with documented proof of cure from HCV may be enrolled), or human immunodeficiency virus (HIV).
12. Subject has a current or recent clinically serious viral, bacterial, fungal, or parasitic infection, including but not limited to the following:

    1. History of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator within 6 months prior to Day 1;
    2. Have active chronic or acute skin infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks prior to Day 1, or superficial skin infections within 1 week prior to Day 1;
    3. History (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster;
    4. Known active tuberculosis (TB) or a positive TB infection test at screening. Subject will be evaluated for latent TB infection with a purified protein derivative (PPD) test or a QuantiFERONTB Gold test. Subjects who demonstrate evidence of latent TB infection (either PPD ≥ 5 mm of induration or positive QuantiFERON-TB Gold test, irrespective of Bacillus Calmette-Guérin vaccination status) will only be allowed to participate in the study if there is documented evidence of a completed adequate treatment course for latent TB (with negative chest x-ray findings for active TB).

    Note: A recent viral upper respiratory tract infection or uncomplicated urinary tract infection should not be considered clinically serious.
13. At screening, any of the following (tests may be repeated once within the same screening period to confirm results prior to Day 1):

    1. Absolute neutrophil count < 1.5 x 109/L;
    2. Absolute lymphocyte count < 0.5 x 109/L;
    3. Hemoglobin < 11.0 g/dL or hematocrit < 30%;
    4. Platelet count < 100 x 109/L;
    5. Clinically significant abnormal estimated creatinine clearance as per investigator judgement (eg, < 90 mL/min based on the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) or serum creatinine value > 1.5 times the upper limit of normal (ULN);
    6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 x the ULN;
    7. Total bilirubin ≥ 1.5 x ULN; subjects with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ≤ ULN.
14. Subject has a history of clinically significant heart disease in the opinion of the investigator (eg, cardiomyopathy, major congenital heart disease, Wolff-Parkinson-White syndrome, heart attack, stroke, or blood clots).
15. Subject is currently receiving anti-coagulants or medications known to cause thrombocytopenia (unless considered safe by the investigator to stop and washout for the duration of the study).
16. Active forms of other inflammatory skin disease(s) or evidence of other skin conditions on the scalp (eg, psoriasis, seborrheic dermatitis, lupus) at screening and/or Day 1, that in the opinion of the investigator might interfere with evaluation of hair regrowth.
17. Subject has presence of any tattoos, scratches, open sores, or skin damages in the target treatment areas that, in the opinion of the investigator, may interfere with study evaluations.
18. Subject is currently treated or was treated within 4 weeks prior to Day 1 with any systemic treatment or oral medication for inflammatory condition; short half-life medications like ibuprofen and paracetamol are acceptable.
19. Subject is currently receiving a nonbiological investigational product or device or has received one within 4 weeks prior to Day 1.
20. Subject has received a live or live-attenuated vaccine within 4 weeks prior to Day 1 or plans to receive a live or live-attenuated vaccine during the study and up to 4 weeks or 5 half-lives (of the study product), whichever is longer, after the last study product administration.
21. Use of systemic and/or intralesional steroids within 8 weeks of Day 1 visit. Note: Intranasal and inhaled corticosteroids are allowed. Eye and ear drops containing corticosteroids are also allowed.
22. Use of systemic treatments including, but not limited to, anthralin, squaric acid, diphenylcycloprophenone (DPCP), dinitrochlorobenzene (DCNB), tacrolimus, minoxidil, or any other medication which in the opinion of the investigator may affect hair regrowth within 4 weeks of Day 1 visit.
23. Subject has received any ultraviolet (UV)-B phototherapy (including tanning beds), has had psoralen-UV-A (PUVA) treatment, or excimer laser within 4 weeks prior to Day 1.
24. Topical medicated treatment that could affect AA including, but not limited to, topical corticosteroids, calcineurin inhibitors, minoxidil, antimicrobials, JAK inhibitors, medical devices within 2 weeks prior to Day 1 visit.

    Note: Topical corticosteroids are permitted outside of the scalp.
25. Subject has previously used a systemic JAK inhibitor for their AA (eg, baricitinib, ritlecitinib, deuruxolitinib) for more than 4 weeks.

    Note: Subjects that used a systemic JAK inhibitor for AA for less than 4 weeks, or used a systemic JAK inhibitor for another reason than AA, are allowed but must have discontinued the systemic JAK inhibitor at least 6 months prior to Day 1.
26. Use of platelet-rich plasma injections in the last 12 weeks prior to Day 1.
27. Subject has received any marketed or investigational biological agent within 12 weeks or 5 half lives (whichever is longer) prior to Day 1.
28. Subject who has had previous treatment with any biologic B-cell-depleting therapy (eg, rituximab, ocrelizumab, or ofatumumab) or other B-cell targeting therapy (eg, belimumab) within 12 months before Day 1.
29. Subject who has received previous treatment with pDC inhibiting therapies (eg, anti immunoglobulin-like transcript [ILT]7, anti-blood dendritic cell antigen 2 [BDCA2]).
30. Subject has a known or suspected allergy to ALD-102 or any component of the investigational product.
31. Subject has a known history of clinically significant drug or alcohol abuse in the last year prior to Day 1.
32. Subject has a history of an allergic reaction or significant sensitivity to lidocaine or other local anesthetics.
33. Subject has a history of hypertrophic scarring or keloid formation in scars or suture sites.
34. Subject has taken anticoagulant medication, such as heparin, low molecular weight (LMW) heparin, warfarin, antiplatelets (except low-dose aspirin ≤ 81 mg which will be allowed), within 2 weeks prior to Day 1, or has a contraindication to skin biopsies. Short half-life nonsteroidal anti-inflammatory drugs (NSAIDs) will not be considered antiplatelets and will be allowed.
35. Subject is not able to tolerate intradermal injection or has a known sensitivity to needle injection.
36. Subject is institutionalized because of legal or regulatory order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse effects (AEs) and severe adverse effects (SAEs) as assessed by CTCAE v5.0, and injection site reactions (ISRs), evaluated by local tolerability assessments and numerical scales. | Daily clinical assessments for 3 days and after 1 week following 1st treatment administration, then approximately every 4 weeks during treatment and follow-up periods for a total of 24 weeks.
  AEs assessed by guidelines outlined in CTCAE v5.0 at baseline, daily for 3 days and after 1 week following the 1st treatment administration, then every 4 weeks during treatment and follow-up periods. ISRs assessed by local tolerability assessments (LTA), including evaluation by the investigator of erythema, swelling/induration, and bruising, and evaluation by the subject of burning/stinging and itching. Grading using a 4-point scale of 0 to 3 (non, mild, moderate, severe) will be used to assess each sign. Pain at each treatment area will also be assessed using a pain numerical rating scale (NRS). Subjects will be asked to assign a numerical score representing the average pain intensity on a scale of 0 to 10, experienced during and after product administration. The LTA and pain assessments will be done approximately 1 & 6h after study product administration at Day 1, Week 4 and Week 8, then after 2 weeks and 6 weeks following last study product administration.

SECONDARY OUTCOMES:
Concentration of ALD-102 in skin biopsies at Week 10 and plasma concentration of ALD-102 over time. | Skin biopsies will be collected at baseline and Week 10. Blood samples will be collected before product administration and approximately 1, 2, 3, 4, 6, and 24 hours after first and last product administration at once at Day 2, Week 1 and Week 16.
  Skin biopsies will be collected to measure drug concentration in skin.
  Blood samples will be collected to measure the systemic exposure of ALD-102 in plasma.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Options Research Group, West Lafayette, Indiana
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (3):
  - The Centre for Clinical Trials, Oakville, Ontario
  - Innovaderm, Montreal, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No